CLINICAL TRIAL: NCT02397642
Title: Dual Trigger Versus Booster Dose of HCG on Ovum Pickup Day in Antagonist IVF/ICSI Cycles Triggered With GnRH Agonist in High Responder Females to Salvage the Luteal Phase
Brief Title: Dual Trigger Versus Booster Dose of HCG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Nile Ivf Center, Cairo, Egypt (Other); Adam International Hospital (Other)
Responsible Party: Principal Investigator, Yasmin Ahmed Bassiouny, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12015
Record Dates: First submitted 2015-03-16; First posted 2015-03-25 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual trigger (Active Comparator): GnRH agonist plus 1000 IU of HCG to trigger final maturation
  Interventions: Procedure: IVF/ICSI; Drug: Human Chorionic Gonadotropin
- Booster HCG dose (Active Comparator): GnRH agonist only to trigger final maturation followed by a booster dose of 1500 IU of HCG on the day of ovum pickup
  Interventions: Procedure: IVF/ICSI; Drug: Human Chorionic Gonadotropin

INTERVENTIONS:
Procedure: IVF/ICSI
Drug: Human Chorionic Gonadotropin — given in different doses and timing to support the luteal phase

SUMMARY:
To salvage the luteal phase and improve pregnancy rate in antagonist IVF/ICSI cycles triggered with GnRH agonist. Two strategies are compared dual trigger with GnRH agonist plus 1000 IU of HCG or triggering with GnRH and giving a booster dose of HCG (1500 IU) on the day of ovum pickup.

ELIGIBILITY:
Inclusion Criteria:

* High responder females undergoing antagonist protocol IVF/ICSI cycle
* More than 14 MII oocytes
* Estradiol more than 3500 pg/ml on day of trigger

Exclusion Criteria:

* Any other protocol
* Normal or poor responders

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 1 year
  The number of cycles with a evidence of a gestational sac with fetal pulstaions after 5 weeks from pregnancy test

SECONDARY OUTCOMES:
OHSS rate | 1 year
  The number of cycles with evidence of OHSS

OTHER OUTCOMES:
Chemical pregnancy rate | 1 year
  The numbr of cycles with a positive pregnancy test after 14 days from embryo transfer
Early miscarriage rate | 1 year
  Pregnancies ending with miscarriage before 12 weeks of gestation
Ongoing pregnancy rate | 1 year
  Pregnancies ongoing beyond 12 weeks of gestation
Live birth rate | 1 year
  Pregnancies ending in a live birth

CONTACTS AND LOCATIONS:
Overall Officials: Sarwat Ahwany, MD, Study Director — Cairo University
Locations (3):
- Egypt (3):
  - IVF centre, Obstetrics and Gynaecology Department, Cairo University Hospitals (Kasr EL Aini), Cairo
  - Adam International hospital, Giza
  - Nile IVF center, Giza